CLINICAL TRIAL: NCT06845696
Title: Comparison of Brugger's Relief Exercises Versus Kinesio Taping at Craniovertebral Angle on Forward Head Posture
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: REC/MS-OMPT/014522 Mahjabeen
Record Dates: First submitted 2025-02-20; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Forward Head Posture
Keywords: Forward head posture; Kinesio taping; Brugger reliefs exercise; Craniovertebral angle

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- kinesiotaping (Experimental): Kinesio taping (KT) is a thin elastic tape which can be stretched up to 130-140% of its original length thereby providing constant shear force on the skin.KT has beneficial effects and possible useful mechanisms to suppress pain, relax muscles, support joints, and improve circulation.Kinesio taping is used for releasing tension on trapezius and erector spinal muscle and to correct the posture.
  Interventions: Other: kinesiotaping
- Bruggers relief exercise (Experimental): Bruegger's postural relief position is an effective self-care exercise for correcting forward head posture. This exercise strengthens the muscles that retract the shoulder blades back while stretching the muscles that protract them forward. By pulling the shoulders back and holding the neck in a chin tuck position, the deep muscles in the neck also become stronger. Bruegger relief exercises (BRE) have been found to be very beneficial for patient rehabilitation
  Interventions: Other: Brugger relief exercise

INTERVENTIONS:
Other: kinesiotaping — Before applying the tape, the treated area was cleaned and shaved. A Y strip of the tape was used to facilitate muscle contraction of the semispinalis capitis with 15 -25% tension in elongated muscle position and three I strip are used in it to release tight upper trapezius, facilitate middle trapezius and to correct posture. 3 days a week for 4 weeks
  Arms: kinesiotaping
Other: Brugger relief exercise — This protocol includes that the patient is positioned on edge of a chair with his hips abducted, feet externally rotated, his head up, his forearms supinated, and wrists and fingers extended. the participants were instructed to perform scapular retraction with chin tucked in, shoulder external rotation, elbow extension, shoulder abduction, and extension. While actively moving their arms and spreading their fingers externally, patient exhaled through lips 12 reps 4 set for 3 days a week Intervention will be given for 4 weeks
  Arms: Bruggers relief exercise

SUMMARY:
The aim of this research is to compare the effect of Brugger relief exercise versus Kinesio taping at craniovertebral angle on forward head posture. Randomized controlled trials done at we care physical therapy clinic Islamabad. The sample size was 28. The subjects were divided in two groups, 14 subjects in Kinesio taping group and 14 in Brugger relief exercise group. Study duration was of 6 months. Sampling technique applied was non probability purposive sampling technique. Only 20-40 years people with forward head posture having craniovertebral angle less than 50° degrees were included. Tools used in the study is protractor app. Data will be analyzed through SPSS 21

DETAILED DESCRIPTION:
Forward head posture (FHP) is a common condition characterized by abnormal cervical spine, leading to non-specific neck pain (NNP). FHP affects millions of people worldwide, causing pain, reduced productivity and quality of life. Current treatments for NNP associated with FHP include exercise programs and Kinesio taping, but there is limited evidence comparing their effectiveness.

The Brugger relief exercises (BRE) consist of a set of exercises designed to target the cervical spine and adjacent muscles with the goal of enhancing posture, alleviating discomfort, and improving functionality. In contrast, Kinesio taping (KT) is a non-invasive and painless method that involves applying gentle traction to the skin, purportedly leading to the reduction of pain and inflammation. This study aims to compare the effectiveness of BRE versus KT on CVA due to FHP. This research will offer important information on the effectiveness of BRE and KT, guiding healthcare providers and patients in selecting the best treatment for FHP-related NNP. The results will support the creation of evidence-backed protocols for addressing FHP-related NNP, ultimately leading to better treatment results and improved quality of life for those affected

ELIGIBILITY:
Inclusion Criteria:

* Both gender
* Patients whose age lies between 20 and 40
* Forward head posture with craniovertebral angle less than 50° degrees

Exclusion Criteria:

* Individuals with pre-existing musculoskeletal conditions affecting posture e.g. scoliosis, Scheuermann's disease.
* Those currently undergoing physical therapy or other posture correction treatments.
* Pregnant individuals, due to potential physiological changes affecting posture.
* Subjects with a history of significant spinal or neck injuries.
* No neurological disease (e.g. cervical radiculopathy, SCI).
* Patients were excluded who shows positive result to spurling test, ULTT, Allen test.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-01-22 (Actual); Primary Completion 2025-09-20 (Estimated); Study Completion 2025-09-20 (Estimated)

PRIMARY OUTCOMES:
CRANIOVERTEBRAL ANGLE | from baseline to 4th week
  This angle is used to assess the forward head posture of the participants. It involves measuring the angle between a horizontal line and a line connecting the C7 vertebrae and the tragus of ear by protractor app.

CONTACTS AND LOCATIONS:
Overall Officials: Asmar Fatima, MS-OMPT, Principal Investigator — Riphah International University
Locations (1):
- We Care Physical Therapy Clinic, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No